CLINICAL TRIAL: NCT00952276
Title: Immunogenicity and Safety of Multiple Formulations of an Adjuvanted A/H1N1 Pandemic Vaccine in Healthy Adult and Elderly Subjects
Brief Title: A Study of Different Formulations of an Adjuvanted A/H1N1 Pandemic Vaccine in Healthy Adults and the Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FUF16; UTN: U1111-1111-4882
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Results first posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-08

CONDITIONS: Influenza; Swine-origin A/H1N1 Influenza
Keywords: Influenza Pandemic Flu Swine-origin A/H1N1 Influenza Adults
MeSH Terms: conditions — Influenza, Human | interventions — Adjuvants, Pharmaceutic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- A/H1N1 Vaccine Group 1 (Experimental): Participants will receive A/H1N1 vaccine formulation 1 (with adjuvant)
  Interventions: Biological: Monovalent Subvirion A/H1N1 influenza vaccine with adjuvant
- A/H1N1 Vaccine Group 2 (Experimental): Participants will receive A/H1N1 vaccine formulation 2 (with adjuvant)
  Interventions: Biological: Monovalent Subvirion A/H1N1 influenza vaccine with adjuvant
- A/H1N1 Vaccine Group 3 (Active Comparator): Participants will receive A/H1N1 vaccine formulation 3
  Interventions: Biological: Monovalent Subvirion A/H1N1 influenza vaccine
- A/H1N1 Vaccine Group 4 (Active Comparator): Participants will receive A/H1N1 vaccine formulation 4
  Interventions: Biological: Monovalent Subvirion A/H1N1 influenza vaccine
- Placebo Group 5 (Placebo Comparator): Participants will receive a placebo vaccine
  Interventions: Biological: Normal saline solution

INTERVENTIONS:
Biological: Monovalent Subvirion A/H1N1 influenza vaccine with adjuvant — 0.5 mL, Intramuscular on Day 0
  Arms: A/H1N1 Vaccine Group 1
Biological: Monovalent Subvirion A/H1N1 influenza vaccine with adjuvant — 0.5 mL, Intramuscular on Day 0
  Arms: A/H1N1 Vaccine Group 2
Biological: Monovalent Subvirion A/H1N1 influenza vaccine — 0.5 mL, Intramuscular on Day 0
  Arms: A/H1N1 Vaccine Group 3
Biological: Monovalent Subvirion A/H1N1 influenza vaccine — 0.5 mL, Intramuscular on Day 0
  Arms: A/H1N1 Vaccine Group 4
Biological: Normal saline solution — 0.5 mL, Intramuscular on Day 0
  Arms: Placebo Group 5

SUMMARY:
The purpose of the study is to evaluate different doses of the Influenza A/H1N1 pandemic vaccine in adults and the elderly.

Primary Objectives:

* To describe the immunogenicity of the candidate vaccines after a single injection.
* To describe the safety of the candidate vaccines after a single injection.

DETAILED DESCRIPTION:
Participants will receive a single injection of their randomized vaccine on Day 0.

ELIGIBILITY:
Inclusion Criteria :

* Healthy adults aged 18 years or older on the day of inclusion
* Informed consent has been signed and dated
* Able to attend all scheduled visits and comply with all trial procedures
* For a woman of child-bearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination, until at least 4 weeks after last vaccination.

Exclusion Criteria :

* Known pregnancy or positive urine pregnancy test
* Currently breastfeeding a child
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination, except for the inactivated seasonal influenza vaccine, within two weeks preceding trial vaccination
* Planned receipt of any vaccine prior to the Day 42 blood sample
* Receipt of blood or blood-derived products in the past 3 months which might interfere with the assessment of immune response
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B antigen, or Hepatitis C
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Self reported thrombocytopenia contraindicating intramuscular (IM) vaccination
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Chronic illness that in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members of the employees or the Investigator
* Previous participation in a swine-origin A/H1N1 pandemic flu trial except if performed in 1976
* Any confirmed case of influenza (including swine-origin A/H1N1 Influenza) since March 2009
* Febrile illness (temperature ≥ 100.4°F [≥ 38.0°C ]) or moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination
* Personal or family history of Guillain-Barré syndrome
* Active neoplastic disease or a history of any hematologic malignancy
* Known seizure/epilepsy history and/or taking anti-seizure medication
* Receipt of psychiatric drugs. Subjects receiving a single antidepressant drug and stable for at least 3 months prior to enrollment, without decompensating symptoms will be allowed to enroll in the study
* Any Grade 1, 2, or 3 liver function values (Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), and Alkaline phosphatase) observed in blood sample taken at Screening
* Any Grade 2 or Grade 3 laboratory abnormalities in blood sample taken at Screening
* Receipt of any monovalent 2009 pandemic H1N1 vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (14):
- United States (14):
  - Anaheim, California
  - Fountain Valley, California
  - South Miami, Florida
  - Springfield, Missouri
  - Rochester, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Grove City, Pennsylvania
  - Jefferson Hills, Pennsylvania
  - Warwick, Rhode Island
  - Jackson, Tennessee
  - Salt Lake City, Utah
  - Springville, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 29 October 2009 to 13 November 2009 at 14 US clinical centers.
Pre-assignment Details: A total of 548 participants who met the inclusion and exclusion criteria were enrolled, vaccinated, and included in data analysis.
Groups:
- Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant: Participants who received a dose of A/H1N1 vaccine containing 3.8 µg hemagglutinin (HA) with adjuvant on Day 0
- Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant: Participants who received a dose of A/H1N1 vaccine containing 7.5 µg hemagglutinin (HA) with adjuvant on Day 0
- Group 3: A/H1N1 Vaccine Formulation 3: Participants who received a dose of A/H1N1 vaccine containing 3.8 µg hemagglutinin (HA) on Day 0
- Group 4: A/H1N1 Vaccine Formulation 4: Participants who received a dose of A/H1N1 vaccine containing 7.5 µg hemagglutinin (HA) on Day 0
- Group 5: Placebo: Participants who received a dose of placebo (normal saline) on Day 0
Period: Overall Study
Arm/Group | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant | Group 3: A/H1N1 Vaccine Formulation 3 | Group 4: A/H1N1 Vaccine Formulation 4 | Group 5: Placebo
Started | 127 | 115 | 122 | 121 | 63
Completed | 126 | 115 | 122 | 120 | 63
Not Completed | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant | Group 3: A/H1N1 Vaccine Formulation 3 | Group 4: A/H1N1 Vaccine Formulation 4 | Group 5: Placebo | Total
Number analyzed (Participants) | 127 | 115 | 122 | 121 | 63 | 548
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 75 | 69 | 73 | 71 | 38 | 326
  >=65 years | 52 | 46 | 49 | 50 | 25 | 222
Age Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 54.0 (18.4) | 53.3 (18.7) | 51.9 (18.0) | 52.7 (19.9) | 54.7 (16.7) | 53.4 (18.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 65 | 66 | 68 | 45 | 323
  Male | 48 | 50 | 56 | 53 | 18 | 225
Region of Enrollment [Number; unit: Participants]
  United States | 127 | 115 | 122 | 121 | 63 | 548

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Detectable Antibodies Before and Following Vaccination With Either Adjuvanted or Non-adjuvanted A/H1N1 Pandemic Vaccine or a Placebo: Age 18 to 64 Years
Description: Antibodies to vaccine were measured using the Hemagglutinin Inhibition (HAI) assay. Detectable anti HA antibody titer was defined as titers ≥ 10 (1/dilution) on Day 0 and Day 21 post-vaccination.
Time Frame: Day 0 and Day 21 post-vaccination
Population: Pre and post-vaccination antibody titers were assessed in the per-protocol population aged 18 to 64 years.
Measure: Number; unit: Participants
Arm/Group | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant | Group 3: A/H1N1 Vaccine Formulation 3 | Group 4: A/H1N1 Vaccine Formulation 4 | Group 5: Placebo
Number analyzed (Participants) | 72 | 67 | 72 | 68 | 38
Participants
  Day 0 (Pre-vaccination) | 44 | 41 | 51 | 46 | 22
  Day 21 (Post-vaccination) | 71 | 67 | 71 | 68 | 27

2. Primary Outcome: Number of Participants With Seroprotection Before and Following Vaccination With Either Adjuvanted or Non-adjuvanted A/H1N1 Pandemic Vaccine or a Placebo: Age 18 to 64 Years
Description: Antibodies to vaccine were measured using the Hemagglutinin Inhibition (HAI) assay. Seroprotection was defined as a titer ≥ 40 (1/dil).
Time Frame: Day 0 and Day 21 post-vaccination
Population: Pre and post-vaccination antibody titers were assessed in the per-protocol population aged 18 to 64 years.
Measure: Number; unit: Participants
Arm/Group | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant | Group 3: A/H1N1 Vaccine Formulation 3 | Group 4: A/H1N1 Vaccine Formulation 4 | Group 5: Placebo
Number analyzed (Participants) | 72 | 67 | 72 | 68 | 38
Participants
  Day 0 (Pre-vaccination) | 25 | 24 | 26 | 27 | 11
  Day 21 (Post-vaccination) | 71 | 66 | 67 | 64 | 13

3. Primary Outcome: Geometric Mean Titers (GMTs) of A/H1N1 Antibodies Before and Following Vaccination With Either Adjuvanted or Non-adjuvanted A/H1N1 Pandemic Vaccine or a Placebo: Age 18 to 64 Years
Description: Antibodies to vaccine were measured using the Hemagglutinin Inhibition (HAI) assay.
Time Frame: Day 0 and Day 21 post-vaccination
Population: Pre and post-vaccination antibody titers were assessed in the per-protocol population aged 18 to 64 years.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant | Group 3: A/H1N1 Vaccine Formulation 3 | Group 4: A/H1N1 Vaccine Formulation 4 | Group 5: Placebo
Number analyzed (Participants) | 72 | 67 | 72 | 68 | 38
Titers
  Day 0 (Pre-vaccination) | 23.7 [16.2 to 34.6] | 21.0 [14.4 to 30.5] | 23.8 [17.1 to 33.1] | 27.7 [18.4 to 41.7] | 20.0 [11.2 to 35.7]
  Day 21 (Post-vaccination) | 896 [673 to 1195] | 900 [653 to 1241] | 470 [314 to 705] | 608 [423 to 875] | 26.3 [15.0 to 46.0]

4. Primary Outcome: Number of Participants With Detectable Antibodies Before and Following Vaccination With Either Adjuvanted or Non-adjuvanted A/H1N1 Pandemic Vaccine or a Placebo: Age ≥ 65 Years
Description: Antibodies to vaccine were measured using the Hemagglutinin Inhibition (HAI) assay. Detectable anti-HA antibody titer was defined as titers ≥ 10 (1/dil).
Time Frame: Day 0 and Day 21 post-vaccination
Population: Pre and post-vaccination antibody titers were assessed in the per-protocol population aged 65 years or older.
Measure: Number; unit: Participants
Arm/Group | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant | Group 3: A/H1N1 Vaccine Formulation 3 | Group 4: A/H1N1 Vaccine Formulation 4 | Group 5: Placebo
Number analyzed (Participants) | 51 | 45 | 47 | 50 | 25
Participants
  Day 0 (Pre-vaccination) | 35 | 39 | 37 | 38 | 19
  Day 21 (Post-vaccination) | 50 | 45 | 46 | 50 | 18

5. Primary Outcome: Number of Participants With Seroprotection Before and Following Vaccination With Either Adjuvanted or Non-adjuvanted A/H1N1 Pandemic Vaccine or a Placebo: Age ≥ 65 Years
Description: as for outcome 2
Time Frame: Day 0 and Day 21 post-vaccination
Population: Pre and post-vaccination antibody titers were assessed in the per-protocol population aged 65 years or older.
Measure: Number; unit: Participants
Arm/Group | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant | Group 3: A/H1N1 Vaccine Formulation 3 | Group 4: A/H1N1 Vaccine Formulation 4 | Group 5: Placebo
Number analyzed (Participants) | 51 | 45 | 47 | 50 | 25
Participants
  Day 0 (Pre-vaccination) | 23 | 21 | 19 | 20 | 9
  Day 21 (Post-vaccination) | 48 | 44 | 40 | 40 | 9

6. Primary Outcome: Geometric Mean Titers (GMTs) of A/H1N1 Antibodies Before and Following Vaccination With Either Adjuvanted or Non-adjuvanted A/H1N1 Pandemic Vaccine or a Placebo: Age ≥ 65 Years
Description: Antibodies to vaccine were measured using the Hemagglutinin Inhibition (HAI) assay.
Time Frame: Day 0 and Day 21 post-vaccination
Population: Pre and post-vaccination antibody titers were assessed in the per-protocol population aged 65 years or older.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant | Group 3: A/H1N1 Vaccine Formulation 3 | Group 4: A/H1N1 Vaccine Formulation 4 | Group 5: Placebo
Number analyzed (Participants) | 51 | 45 | 47 | 50 | 25
Titers
  Day 0 (Pre-vaccination) | 28.5 [18.3 to 44.3] | 40.0 [25.7 to 62.2] | 26.1 [18.3 to 37.2] | 23.0 [16.4 to 32.1] | 25.7 [14.6 to 45.2]
  Day 21 (Post-vaccination) | 501 [330 to 761] | 630 [432 to 920] | 177 [108 to 292] | 189 [118 to 301] | 26.8 [14.7 to 48.8]

7. Primary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reaction Following Vaccination With Either Adjuvanted or Non-adjuvanted A/H1N1 Pandemic Vaccine or a Placebo: Age 18 to 64 Years
Description: Solicited Injections Site Reactions: Pain, Erythema, Swelling, Induration, and Ecchymosis. Solicited Systemic Reactions: Fever (Temperature), Headache, Malaise, Myalgia, and Shivering
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent to treat population aged 18 to 64 years.
Measure: Number; unit: Participants
Arm/Group | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant | Group 3: A/H1N1 Vaccine Formulation 3 | Group 4: A/H1N1 Vaccine Formulation 4 | Group 5: Placebo
Number analyzed (Participants) | 75 | 69 | 73 | 71 | 38
Participants
  Any Solicited Injection Site Pain | 52 | 53 | 13 | 17 | 11
  Grade 3 Pain (Prevents daily activity) | 1 | 2 | 1 | 0 | 0
  Any Solicited Injection Site Erythema | 2 | 2 | 2 | 0 | 0
  Grade 3 Erythema (> 10 cm) | 0 | 0 | 0 | 0 | 0
  Any Solicited Injection Site Swelling | 3 | 1 | 0 | 0 | 0
  Grade 3 Swelling (> 10 cm) | 0 | 0 | 0 | 0 | 0
  Any Solicited Injection Site Induration | 1 | 3 | 0 | 0 | 0
  Grade 3 Induration (> 10 cm) | 0 | 0 | 0 | 0 | 0
  Any Solicited Injection Site Ecchymosis | 4 | 0 | 1 | 0 | 0
  Grade 3 Ecchymosis | 0 | 0 | 0 | 0 | 0
  Any Fever | 1 | 0 | 3 | 0 | 0
  Grade 3 Fever (≥ 102.1 ºF or ≥ 39.0 ºC) | 0 | 0 | 0 | 0 | 0
  Any Headache | 36 | 27 | 25 | 24 | 15
  Grade 3 Headache (Prevents daily activity) | 2 | 3 | 1 | 0 | 0
  Any Malaise | 29 | 21 | 20 | 12 | 8
  Grade 3 Malaise (Prevents daily activity) | 3 | 3 | 3 | 2 | 0
  Any Myalgia | 36 | 28 | 12 | 17 | 12
  Grade 3 Myalgia (Prevents daily activity) | 3 | 4 | 3 | 2 | 0
  Any Shivering | 6 | 7 | 6 | 6 | 3
  Grade 3 Shivering (Prevents daily activity) | 1 | 2 | 1 | 0 | 0

8. Primary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reaction Following Vaccination With Either Adjuvanted or Non-adjuvanted A/H1N1 Pandemic Vaccine or a Placebo: Age ≥ 65 Years
Description: as for outcome 7
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population aged 65 years or older.
Measure: Number; unit: Participants
Arm/Group | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant | Group 3: A/H1N1 Vaccine Formulation 3 | Group 4: A/H1N1 Vaccine Formulation 4 | Group 5: Placebo
Number analyzed (Participants) | 52 | 46 | 49 | 50 | 25
Participants
  Any Solicited Injection Site Pain | 21 | 22 | 2 | 7 | 2
  Grade 3 Pain (Prevents daily activities) | 0 | 1 | 0 | 0 | 0
  Any Solicited Injection Site Erythema | 1 | 1 | 0 | 1 | 0
  Grade 3 Erythema (> 10 cm) | 0 | 0 | 0 | 0 | 0
  Any Solicited Injection Site Swelling | 0 | 3 | 0 | 0 | 0
  Grade 3 Swelling (> 10 cm) | 0 | 0 | 0 | 0 | 0
  Any Solicited Injection Site Induration | 2 | 2 | 0 | 0 | 0
  Grade 3 Induration (> 10 cm) | 0 | 0 | 0 | 0 | 0
  Any Solicited Injection Site Ecchymosis | 0 | 0 | 0 | 2 | 1
  Grade 3 Ecchymosis (> 10 cm) | 0 | 0 | 0 | 0 | 0
  Any Fever | 0 | 1 | 0 | 1 | 0
  Grade 3 Fever (≥ 102.1 ºF or ≥ 39.0 ºC) | 0 | 0 | 0 | 0 | 0
  Any Headache | 10 | 10 | 5 | 10 | 3
  Grade 3 Headache (Prevents daily activity) | 2 | 1 | 0 | 0 | 0
  Any Malaise | 8 | 4 | 3 | 5 | 1
  Grade 3 Malaise (Prevents daily activity) | 0 | 0 | 0 | 1 | 0
  Any Myalgia | 12 | 11 | 3 | 7 | 2
  Grade 3 Myalgia (Prevents daily activity) | 1 | 1 | 0 | 0 | 0
  Any Shivering | 2 | 3 | 1 | 3 | 1
  Grade 3 Shivering (Prevents daily activity) | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination (Day 0) up to 12 months post-vaccination.
Arm/Group | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant | Group 3: A/H1N1 Vaccine Formulation 3 | Group 4: A/H1N1 Vaccine Formulation 4 | Group 5: Placebo
Serious Adverse Events (participants affected / at risk) | 6/127 | 5/115 | 5/122 | 4/121 | 5/63
Other Adverse Events (participants affected / at risk) | 77/127 | 75/115 | 75/122 | 82/121 | 40/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant (N=127) | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant (N=115) | Group 3: A/H1N1 Vaccine Formulation 3 (N=122) | Group 4: A/H1N1 Vaccine Formulation 4 (N=121) | Group 5: Placebo (N=63)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: A/H1N1 Vaccine Formulation 1 + Adjuvant (N=127) | Group 2: A/H1N1 Vaccine Formulation 2 + Adjuvant (N=115) | Group 3: A/H1N1 Vaccine Formulation 3 (N=122) | Group 4: A/H1N1 Vaccine Formulation 4 (N=121) | Group 5: Placebo (N=63)
Injection site pain (General disorders) | 73 (73) | 75 (75) | 15 (15) | 24 (24) | 13 (13)
Malaise (General disorders) | 37 (37) | 25 (25) | 23 (23) | 17 (17) | 9 (9)
Shivering (General disorders) | 8 (8) | 10 (10) | 7 (7) | 9 (9) | 4 (4)
Haemoglobin decreased (Investigations) | 77 (90) | 70 (78) | 69 (77) | 81 (91) | 37 (42)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 10 (10) | 7 (7) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 48 (48) | 39 (39) | 15/121 (15) | 14 (14) | 14 (14)
Headache (Nervous system disorders) | 46 (46) | 37 (37) | 30 (30) | 34 (34) | 18 (18)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (8) | 2 (2) | 6 (7) | 2 (2)
Headache (Nervous system disorders) | 7 (10) | 6 (6) | 6 (12) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.